CLINICAL TRIAL: NCT03453216
Title: Impact of the Presence of a Familiar Peer of the Same Age on the Behavioral Performance of the Child, Adolescent, and Young Adult and Study of the Biological Correlates by Neuroimagery
Brief Title: Impact of Another Person's Presence on Brain and Behavioral Performance
Acronym: SOFEE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator Departure
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-A01477-44
Record Dates: First submitted 2018-02-14; First posted 2018-03-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Behavior and Behavior Mechanisms
MeSH Terms: conditions — Behavior | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral test and fMRI (Experimental): Neuropsychological tests and training in behavioral tasks and a Functional Magnetic Resonance Imaging (fMRI) exam
  Interventions: Behavioral: neuropsychological tests

INTERVENTIONS:
Behavioral: neuropsychological tests — Part 1: to determine the cognitive capacity, the subjects undergo different neuropsychological tests To determine individual characteristics children, adolescents and adults complete self-assessment questionnaires .
  Adults spend a semi-directive interview. Part 2: while the subject 1 (S1) is installed in the MRI, he perform behavioral tasks with the subject 2 (S2) (familiar peer of the same age ± 2 years) installed in an adjacent room, alternating periods when S1 is observed by S2 (condition "Social") and periods when S1 is not observed by S2 (condition "Alone").
  Other Names: Functional Magnetic Resonance Imaging (fMRI) exam

SUMMARY:
In a recent study, investigators provided the first neuroscientific data on social facilitation. This neuroimaging study, performed in the macaque monkey, shows a marked improvement in performance in a simple task when a congener is present compared to when the animal performs the task alone. This social facilitation is accompanied by a significant increase in brain activity within the fronto-parietal network of attention. No variation in activity, however, is observed in the cerebral network of motivation. These results argue in favor of the implication of attentional processes in the phenomenon of social facilitation. The challenge now is to determine whether social facilitation is always based on the attention network (whatever the task) or, alternatively, whether it increases activity in any cerebral circuit involved depending on the task performed and the population studied. This hypothesis, which the investigators have named the "multi-mediator model of social facilitation", has the advantage of reconciling the attentional and motivational theories of social facilitation, which are not mutually exclusive. This hypothesis also provides an explanation for the pervasiveness (across species and different ages for humans) of social facilitation. The main objective of SOFEE is to gather neuroscientific evidence to support the multi-facilitator model of social facilitation.

DETAILED DESCRIPTION:
The main objective is to study the effect of the presence of others on cognitive performance and its evolution during development by behavioral and neural measures. The secondary objective is to identify factors (psychological characteristics such as personality traits) explaining individual, behavioral and neural differences, sensitivity to the presence of others.

ELIGIBILITY:
Inclusion Criteria:

* Girl or boy aged ≥ 8 years and ≤ 12 years old for children,
* Girl or boy aged ≥ 13 years and ≤ 19 years old for teenagers,
* Woman or man age ≥ 20 years and ≤ 35 years old for young adults,
* French mother tongue,
* With the right to a social security scheme or similar,
* With informed consent form signed by the legal representatives and the subject, for minors,
* Has signed the informed consent form, for adults.

Exclusion Criteria:

* Known acquired neurological disorders, including epilepsy,
* Known psychiatric disorders,
* Complications at birth requiring admission to neonatal intensive care unit,
* Ongoing treatment with drugs affecting the central nervous system,
* Significant hearing impairment,
* Uncorrected visual inadequacy,
* Left manual preference,
* Contraindications to the MRI examination (people using a pacemaker or an insulin pump, people wearing a metal prosthesis or an intracerebral clip as well as claustrophobic subjects),
* Refusal of the subject or parents of the subject to be informed of any anomalies detected on the MRI,
* Pregnancy for women of childbearing age: the possibility of pregnancy will be ruled out on questioning for inclusion,
* Protected persons other than children

Ages: 8 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 112 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Behavioral performance evaluation | an average of 5 years
  percentage of correct answers and reaction time when performing cognitive number and rhyme comparison tasks in the presence or absence of a familiar peer
identification through Functional Magnetic Resonance Imaging (fMRI ) of brain activity related to the presence of others | an average of 5 years
  Comparison of activity in the three populations tested (children, adolescents, adults)

SECONDARY OUTCOMES:
Determination of individual characteristics | an average of 5 years
  answers of self-assessment questionnaires and semi-directive interview

CONTACTS AND LOCATIONS:
Overall Officials: POISSON ALICE, MD, Principal Investigator — CH LE VINATIER
Locations (1):
- CH Le Vinatier, Bron, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: Undecided